CLINICAL TRIAL: NCT05344898
Title: Subscapularis Repair in Reverse Shoulder Arthroplasty: A Multi-Center Randomized Single Blinded Superiority Study
Brief Title: Subscap Reverse Shoulder Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mohit N. Gilotra, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00100825
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Injuries; Rotator Cuff Injuries
MeSH Terms: conditions — Shoulder Injuries; Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subscap Tenotomy (Experimental): The subscapularis tendon is not repaired.
  Interventions: Procedure: Subscap Tenotomy
- Subscap Repair (Experimental): The subscapularis tendon is repaired.
  Interventions: Procedure: Subscap Repair

INTERVENTIONS:
Procedure: Subscap Tenotomy — Group will not have their subscapularis tendon repaired following a reverse shoulder replacement.
  Arms: Subscap Tenotomy
Procedure: Subscap Repair — Group will have their subscapularis tendon repaired following a reverse shoulder replacement.
  Arms: Subscap Repair

SUMMARY:
The subscapularis is part of the rotator cuff and is release as part of a reverse shoulder replacement. The decision to repair this tendon is controversial. This research is being done to help determine if rotator cuff repair improves or hinders shoulder replacement. A worrisome but rare complication after shoulder replacement is dislocation. Rotator cuff repair may help reduce this risk. The repair may hinder some of the range of motion afterwards or could help with internal rotation strength. There is a chance that the repair doesn't matter at all. The goal of this study is to delineate outcomes after reverse shoulder arthroplasty with the respect to management of the subscapularis tendon. Further information about rotator cuff repair after reverse shoulder replacement can help define complications, potentially decrease OR time, and improve functional outcomes. A total of 148 patients will be enrolled and the duration of the study will be 5 years. All patients will be required to follow-up at 2¬-week, 6-week, 3-month, 6-month, 1-year, and 2-year post-operative marks. Any time information is collected for a study there is a small risk of breach of confidentiality. There are no monetary costs or payments associated with this study. You may or may not benefit by taking part in this study. There is no guarantee that you will receive direct benefit from your participation in this study. To be clear, participation in this study is completely voluntary.

DETAILED DESCRIPTION:
You're going to undergo a procedure called a reverse shoulder replacement and I'm sure Dr. Gilotra already went over the procedure with you but I will again briefly. Before the hardware is put in, there is a tendon in your shoulder that has to be "released". It's released because the doctor has to move it out of the way to get to your shoulder joint. Now when the hardware has been implanted and the surgery is complete, the doctor now has two options. He can decide to repair this tendon or not. The thing is due to the hardware that is implanted, your shoulder doesn't really need this tendon anymore to help it move. So, there are some doctors in the country who choose to repair the tendon and there are some doctors who choose to just let it be. Patients have done great with either or.

We are performing this nationwide study to see if one option (between repairing this tendon or leaving it) is slightly better than the other. There is a chance that repairing the tendon can decrease the risk of dislocations in the future and also help you move your arm better. There is a chance that this repair doesn't matter at all. If we figure out whether to repair or not to repair this tendon, we will be able to better define complications, potentially decrease surgery time, and improve how well patients perform daily activities.

We randomize you to the repair on don't repair group, almost like flipping a coin. With me, you'll be answering simple questions that will track your functionality over time.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 95 years old
2. Undergoing reverse shoulder arthroplasty for any indication including revision surgery

Exclusion Criteria:

1. Irreparable Subscapularis Tendon

   a. Reparability of Subscapularis will be determined based on MRI or CT scan obtained preoperatively and confirmed intraoperatively. Tendons must be intact with less than Grade I or II Fatty Infiltration as determined by the Goutallier classification.
2. Any history of proximal humerus fracture
3. Any revision with proximal humerus bone loss

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in Internal Rotation | Pre-op and post-op Months 3,6,12,24
  Internal rotation behind the back
Change in BOSS Scores | Pre-op and post-op Months 3,6,12,24
  Change in Baltimore Orthopaedic Subscapularis Score (BOSS) over 2 years. The score asks enrolled patients a series of questions. The answer choices are the following: No difficulty, mild difficulty, severe difficulty, unable to perform.

SECONDARY OUTCOMES:
Change in ASES score | Pre-op and post-op Months 3,6,12,24
  Change in American Shoulder and Elbow Surgeon (ASES) score over 2 years postoperatively compared to preoperative. The score ranges from 0 to 10 with 0 indicating no pain and 10 indicating worst pain possible.

OTHER OUTCOMES:
Ultrasound Evaluation | Month 6
  Blinded ultrasound evaluation of subscapularis integrity at 6 months. The "Sugaya classification" will be used to assess the subscapularis integrity. The score ranges from Type 1 to Type 5.
  Type 1: indicating sufficient thickness with homogeneously low intensity
  Type 2: sufficient thickness with partial high intensity
  Type 3: insufficient thickness without discontinuity
  Type 4: the presence of a minor discontinuity
  Type 5: the presence of a major discontinuity

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Gilotra, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otto RJ, Clark RE, Frankle MA. Reverse shoulder arthroplasty in patients younger than 55 years: 2- to 12-year follow-up. J Shoulder Elbow Surg. 2017 May;26(5):792-797. doi: 10.1016/j.jse.2016.09.051. Epub 2016 Dec 26. PMID 28034540
- [Background] Friedman RJ, Flurin PH, Wright TW, Zuckerman JD, Roche CP. Comparison of reverse total shoulder arthroplasty outcomes with and without subscapularis repair. J Shoulder Elbow Surg. 2017 Apr;26(4):662-668. doi: 10.1016/j.jse.2016.09.027. Epub 2016 Oct 27. PMID 28277259
- [Background] Villacis D, Sivasundaram L, Pannell WC, Heckmann N, Omid R, Hatch GF 3rd. Complication rate and implant survival for reverse shoulder arthroplasty versus total shoulder arthroplasty: results during the initial 2 years. J Shoulder Elbow Surg. 2016 Jun;25(6):927-35. doi: 10.1016/j.jse.2015.10.012. Epub 2016 Jan 18. PMID 26796602
- [Background] Vourazeris JD, Wright TW, Struk AM, King JJ, Farmer KW. Primary reverse total shoulder arthroplasty outcomes in patients with subscapularis repair versus tenotomy. J Shoulder Elbow Surg. 2017 Mar;26(3):450-457. doi: 10.1016/j.jse.2016.09.017. Epub 2016 Oct 14. PMID 27751722
- [Background] Kohan EM, Chalmers PN, Salazar D, Keener JD, Yamaguchi K, Chamberlain AM. Dislocation following reverse total shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Jul;26(7):1238-1245. doi: 10.1016/j.jse.2016.12.073. Epub 2017 Feb 3. PMID 28162886
- [Background] Pastor MF, Kraemer M, Wellmann M, Hurschler C, Smith T. Anterior stability of the reverse shoulder arthroplasty depending on implant configuration and rotator cuff condition. Arch Orthop Trauma Surg. 2016 Nov;136(11):1513-1519. doi: 10.1007/s00402-016-2560-3. Epub 2016 Aug 26. PMID 27566617
- [Background] Padegimas EM, Zmistowski BM, Restrepo C, Abboud JA, Lazarus MD, Ramsey ML, Williams GR, Namdari S. Instability After Reverse Total Shoulder Arthroplasty: Which Patients Dislocate? Am J Orthop (Belle Mead NJ). 2016 Nov/Dec;45(7):E444-E450. PMID 28005111
- [Background] Farrington CP, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Stat Med. 1990 Dec;9(12):1447-54. doi: 10.1002/sim.4780091208. PMID 2281232
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518